CLINICAL TRIAL: NCT04252534
Title: Management of Retinitis Pigmentosa Via Repetitive Electromagnetic Stimulation and Autologous Platelet Rich Plasma
Brief Title: Management of Retinitis Pigmentosa Via Electromagnetic Stimulation and Platelet Rich Plasma
Acronym: rEMS
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Ankara Universitesi Teknokent (Other)
Responsible Party: Principal Investigator, Umut Arslan, Principle investigator, MD, Ankara Universitesi Teknokent
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 19-1293-18
Record Dates: First submitted 2020-01-31; First posted 2020-02-05 (Actual); Last update posted 2020-02-05 (Actual); Status verified 2020-02

CONDITIONS: Retinitis Pigmentosa
Keywords: Retinitis pigmentosa; Electromagnetic stimulation; Platelet rich plasma; Magnovision; Ellipsoid zone
MeSH Terms: conditions — Retinitis Pigmentosa

STUDY DESIGN:
Intervention Model Description: Comparative, open label
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Repetitive electromagnetic stimulation (Active Comparator): Group 1 consists of 20 RP patients (40 eyes) who received combined rEMS with PRP. In this group, patients received rEMS for 30 minutes before subtenon PRP injections. In this group, 3 loading doses were applied at 3-week intervals. Then 2 booster dose were applied at 6-month intervals.
  Interventions: Combination Product: PRP combined Magnovision; Biological: PRP
- Platelet rich plasma (Active Comparator): Group 2 consists of 20 RP patients (40 eyes). In this group, patients received only subtenon PRP injections. In this group, 3 loading doses were applied at 3-week intervals. Then 2 booster dose were applied at 6-month intervals.
  Interventions: Biological: PRP
- Natural course (No Intervention): Group 3 consists of 20 RP patients (40 eyes). Patients in this group did not accept any interventional application and were only followed up. The

INTERVENTIONS:
Combination Product: PRP combined Magnovision — The rEMS helmet is used to stimulate the retina and visual pathways. (MagnovisionTM) combined with subtenon platelet rich plasma injection
  Arms: Repetitive electromagnetic stimulation
Biological: PRP — Fresh autologous platelet rich plasma, injected subtenon space.
  Arms: Platelet rich plasma; Repetitive electromagnetic stimulation

SUMMARY:
The aim of this study is to investigate whether natural progression rate can be slowed down with subtenon PRP or PRP application combined with rEMS in retinitis pigmentosa cases.

DETAILED DESCRIPTION:
Retinitis pigmentosa (RP) is a progressive external retinal degeneration resulting from mutation in any of the 260 genes found in the retinal pigment epithelium (RPE). The progression rate and findings of the disease are heterogeneous according to genetic mutation and heredity type. The initial symptom of the disease is usually night blindness (nyctalopia) beginning in childhood or adolescent period. Narrowing in the visual field and legal blindness develops as the disease progresses. If low grade inflammation is added, the disease is complicated by cataracts, epiretinal membrane and macular edema. In the fundus examination, the appearance of midperiferal bone spicule pigmentation is usually sufficient to diagnosis. Developments in optical coherence tomography (OCT) technology enable detailed imaging of the sensorial retina and the ellipsoid zone. The ellipsoid zone (EZ) is an image of the inner and outer segments of photoreceptor cells. Loss of EZ is considered the gold standard in the diagnosis and follow-up of RP. Visual field monitoring and electroretinography (ERG) are indirect signs of EZ loss and correlated with EZ width. Mutations in RPE disrupt the synthesis of some vital peptide and growth factors for photoreceptors.

Platelet-rich plasma (PRP) is a good source of growth factors. Platelets have more than 30 growth factors and cytokines in α-granules such as neurotrophic growth factor (NGF), neural factor (NF), brain derived neurotrophic factor (BDNF), basic fibroblast growth factor (bFGF), insulin-like growth factor (IGF), transforming growth factor (TGF-β), vascular endothelial growth factor (VEGF), platelet derived growth factor (PDGF) etc. These peptides regulate the energy cycle at the cellular level, local capillary blood flow, neurogenesis and cellular metabolism. Anti-inflammatory effects of PRP are also associated with soluble cytokines.

Repetitive electromagnetic stimulation (rEMS), increases binding affinity and the synthesis of growth factor receptors on neural tissues. It provides electromagnetic iontophoresis by changing the electrical charges of tyrosine kinase receptors (Trk). rEMS forms hyperpolarization-depolarization waves in neurons, thereby increasing neurotransmission and capillary blood flow. Trk receptors are commonly found around limbus, extraocular muscle insertions and the optic nerve. Molecules smaller than 75 kD can pass from the sclera passively to the suprachoroidal space. Electrical or electromagnetic iontophoresis is required for molecules larger than 75kD such as BDNF and IGF to pass through the sclera.

The aim of this study is to investigate whether natural progression rate can be slowed down with subtenon PRP or PRP application combined with rEMS in retinitis pigmentosa cases.

ELIGIBILITY:
Inclusion Criteria:

* RP patients in any phenotype with vision over 50 letters

Exclusion Criteria:

* Media opacity and nystagmus presence to prevent EZW imaging in OCT

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 60 (Actual)
Dates: Start 2017-01-01 (Actual); Primary Completion 2019-12-30 (Actual); Study Completion 2019-12-30 (Actual)

PRIMARY OUTCOMES:
Ellipsoid zone width (EZW) | Change from baseline EZW at 12 months
  The ellipsoid zone (EZ) is an image of the inner and outer segments of photoreceptor cells on OCT view

CONTACTS AND LOCATIONS:
Overall Officials: Umut Arslan, MD, Principal Investigator — Ankara Universitesi Teknokent

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Arslan U, Ozmert E, Demirel S, Ornek F, Sermet F. Effects of subtenon-injected autologous platelet-rich plasma on visual functions in eyes with retinitis pigmentosa: preliminary clinical results. Graefes Arch Clin Exp Ophthalmol. 2018 May;256(5):893-908. doi: 10.1007/s00417-018-3953-5. Epub 2018 Mar 15. PMID 29546474
- [Background] Ozmert E, Arslan U. Management of Deep Retinal Capillary Ischemia by Electromagnetic Stimulation and Platelet-Rich Plasma: Preliminary Clinical Results. Adv Ther. 2019 Sep;36(9):2273-2286. doi: 10.1007/s12325-019-01040-2. Epub 2019 Aug 5. PMID 31385285
- [Background] Ozmert E, Arslan U. Management of retinitis pigmentosa by Wharton's jelly derived mesenchymal stem cells: preliminary clinical results. Stem Cell Res Ther. 2020 Jan 13;11(1):25. doi: 10.1186/s13287-020-1549-6. PMID 31931872
- [Derived] Arslan U, Ozmert E. Management of Retinitis Pigmentosa via Platelet-Rich Plasma or Combination with Electromagnetic Stimulation: Retrospective Analysis of 1-Year Results. Adv Ther. 2020 May;37(5):2390-2412. doi: 10.1007/s12325-020-01308-y. Epub 2020 Apr 18. PMID 32303913